CLINICAL TRIAL: NCT03505047
Title: Immediate Versus Delayed Insertion of the Copper IUD After Second-trimester Medical Abortion - a Randomised Controlled Trial.
Brief Title: Immediate Versus Delayed IUD Insertion After Second Trimester Medical Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Deborah Constant, Dr, Senior Researcher, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 007/2018
Record Dates: First submitted 2018-04-12; First posted 2018-04-23 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Contraception
Keywords: second trimester medical abortion; Immediate versus delayed insertion; copper intrauterine device
MeSH Terms: interventions — Intrauterine Devices, Copper

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate group: (Experimental): The Copper Intrauterine device will be inserted within 24 hours of the expulsion of the fetus and placenta or after surgical evacuation for placental remains, and prior to discharge from the facility.
  Interventions: Device: Copper Intrauterine device
- Delayed Group (No Intervention): The Copper Intrauterine device will be inserted at a local community health centre 14-28 days after discharge.

INTERVENTIONS:
Device: Copper Intrauterine device — Immediate insertion of the copper intrauterine device after completion of abortion
  Arms: Immediate group:

SUMMARY:
The main objective of the study is to compare use, in a randomised controlled trial, of the the copper IUD if inserted immediately after completion of a second trimester medical abortion, to standard care with insertion 3-4 or more weeks after abortion at community health centres.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak English, Afrikaans or Xhosa;
* Requesting and eligible for abortion according to standard practice at the hospital;
* Gestational age 13-20 weeks verified by ultrasound;
* Interested and eligible for the copper IUD as a post-abortion contraceptive method;
* Willingness to participate in the trial including follow-up;
* Able to provide a working phone & telephone number to allow for contact;
* Willing and able to provide informed consent
* Staying within one hour travel time of GSH

Exclusion Criteria:

* Active pelvic inflammatory disease, pelvic tuberculosis; severe thrombocytopenia;
* Positive N. Gonorrhea or C. Trachomatis that has not been adequately treated
* Copper allergy
* Hb <10g/dL
* Uterine anomaly preventing placement of the IUD; cervical cancer or carcinoma in-situ, untreated high grade squamous intraepithelial lesions
* Hemorrhage; or ruptured uterus
* History of ectopic pregnancy
* Wilsons' disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Use of the copper IUD | 6 weeks after second trimester abortion
  Number of women using the IUD
Insertion of the IUD | 6 weeks after second trimester abortion
  Number of IUD insertions

SECONDARY OUTCOMES:
Use of the IUD at 3 months post-abortion | 3 months after second trimester medical abortion
  Number of women using the IUD
Use of the IUD at 6 months post-abortion | 6 months after second trimester medical abortion
  Number of women using the IUD
Spontaneous expulsion of the IUD | 6 weeks post-abortion
  Number of full and partial expulsions
Spontaneous expulsion of the IUD | Between 6 weeks and 3 months post abortion
  Number of full and partial expulsions
Spontaneous expulsion of the IUD | Between 3 and 6 months post abortion
  Number of full and partial expulsions
Removal of IUD and associated factors | within 3 and 6 months post-abortion
  Number of removals
Abortion-related and IUD-related complications | within 3 months post-abortion
  Number of complications
Women's satisfaction and acceptability of the IUD | Reported at 3 and 6 months post-abortion
  5 point scales
Recurrent pregnancy | At 6 months post-abortion
  Number of recurrent pregnancies

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Constant, PhD, Principal Investigator — University of Cape Town
Locations (1):
- Groote Schuur Hospital, Cape Town, Western Province, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Participant data will be made available from an institutional repository
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available following successful publication of findings - Expected date December 2020. No cut-off date
Access Criteria: Through application to lead investigator